CLINICAL TRIAL: NCT02528240
Title: Endodontic Microsurgery With the Use of L-PRF and an Occlusive Membrane: a Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: S58015 / B322201525314/ I / U
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Periapical Periodontitis
Keywords: platelets
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- + L-PRF (Experimental): With leukocyte and platelet rich fibrin
  Interventions: Procedure: EMS; Device: + occlusive membrane; Device: conebeam CT
- - L-PRF (Active Comparator): Without leukocyte and platelet rich fibrin
  Interventions: Procedure: EMS; Device: conebeam CT

INTERVENTIONS:
Procedure: EMS
Device: + occlusive membrane
  Arms: + L-PRF
Device: conebeam CT

SUMMARY:
This study evaluates the effect of leucocyte and platelet rich fibrin (L-PRF) during endodontic microsurgery (EMS) on patient's post-operative comfort and periapical bone healing. Also the influence of an occlusive membrane barrier in EMS on the periapical bone healing will be studied. The trial design is an open randomized controlled clinical trial with a 2x2 factorial design. Half of the participants will receive EMS with L-PRF (experimental group), the other half without (control group). The control and experimental group will be divided in 2 subsequent groups: half of the participants will receive an occlusive membrane during EMS, the other half not.

ELIGIBILITY:
Inclusion Criteria:

* Provision of Informed Consent
* Patients in need of an EMS
* EMS is the only option to cure the periapical lesion

Exclusion Criteria:

* Unlikely to be able to comply with the study procedures, as judged by the investigator
* Orthograde endodontic (re)treatment is indicated
* Known or suspected current malignancy
* History of chemotherapy within 5 years prior to study
* History of radiation in the head and neck region
* History of other metabolic bone diseases
* History of bleeding disorders
* HIV disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Patient related outcomes | 7 days
  Assessed with a Visual Analog Scale

SECONDARY OUTCOMES:
Patient related outcomes | 7 days
  Assessed with a questionnaire

OTHER OUTCOMES:
Amount of periapical bone healing in time | 4 years
  Assessed with conebeam CT and periapical radiography
Timeframe in which the cortical bone plate closes | 1 year
  Assessed with echography
Bone or scar tissue healing | 4 years
  Assessed with conebeam CT
Dentinal defects | 1 day
  Assessed with a LED light source
Type of periapical tissue | 7 days
  Assessed by biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium